CLINICAL TRIAL: NCT02607085
Title: REal World EVidence for TrEAtment of HyperkaLemia in the Emergency Department (REVEAL - ED): a Multicenter, Prospective, Observational Study
Brief Title: REal World EVidence for TrEAtment of HyperkaLemia in Emergency Department: Multicenter, Prospective, Observational Study
Acronym: REVEAL-ED
Status: Completed | Type: Observational
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZS-007
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the management of subjects with Standard of Care (SOC) when admitted to the Emergency Department (ED) with hyperkalemia (potassium value ≥ 5.5 mmol/L). Demographics and medical history data, including previous ED visits and/or hospital admissions for hyperkalemia and reason for current ED admission, will be recorded. Subjects who receive an intervention/treatment for hyperkalemia will have study-related potassium values determined at 30 minutes, 1, 2, and 4 hours after the start of treatment. Subjects who receive no intervention/treatment during the initial 4-hour period will have a study-related potassium value determined 4 hours after the baseline potassium measurement. Available data obtained as part of SOC management will include physical examinations, vital signs, fluid intake and urine output, ECGs, clinical laboratory data, and results of chest x-rays. Data regarding the subject's chief complaint upon admission to the ED, the possible cause of the subject's hyperkalemia, and admitting and discharge diagnosis will be recorded; the subject's overall discharge summary will also be collected.

DETAILED DESCRIPTION:
This study evaluates the management of subjects with Standard of Care (SOC) when admitted to the Emergency Department (ED) with hyperkalemia (potassium value ≥ 5.5 mmol/L). If the initial SOC potassium value is suspect, a second confirmatory SOC sample should be obtained and must be ≥ 5.5 mmol/L to continue study participation. It is acceptable for the site to use a point of care analyzer to obtain SOC potassium if this is the ED's standard practice. Demographics and medical history data, including previous ED visits and/or hospital admissions for hyperkalemia and reason for current ED admission, will be recorded. If a baseline study-related potassium value determined prior to the first intervention/treatment is unable to be obtained, the SOC potassium value that qualified the subject for entry into the study will be used as the subject's baseline. Enrollment of subjects with baseline potassium values < 6.0 mmol/L will be limited to a maximum of 50 subjects.

Subjects who receive an intervention/treatment for hyperkalemia (eg, intravenous [IV] calcium, insulin/glucose, beta2-agonists, diuretics, IV bicarbonate, sodium polystyrene sulfonate (SPS), dialysis and/or other intervention for hyperkalemia) will have study-related potassium values drawn at 30 minutes, 1, 2, and 4 hours after the start of treatment. Subjects who receive no intervention/treatment during the initial 4-hour period will have a study-related potassium value drawn 4 hours after the baseline potassium measurement.

The timing of each intervention/treatment and the collection of recordable outcomes following admission to the ED will be recorded, together with the procedure followed, as well as dose and route of administration. In addition concomitant medications will be collected from 14 days prior to ED admission and will continue until discharge from the ED. If the subject is admitted into other care (eg, hospital, ICU, observational unit, etc), post-ED concomitant medication collection will be performed for up to 7 days following admission to that unit or until discharge from that unit, if earlier.

Recordable outcomes will be limited to pulmonary edema, ventricular tachycardia/fibrillation, pulseless electrical activity arrest, new clinically significant electrocardiogram (ECG) changes (including but not limited to severe bradycardia, advanced heart block, bundle branch block, tachycardia [>100 bpm]), palpitations, hypoglycemia, and gastrointestinal-related events (eg, nausea, vomiting, diarrhea) and any other event deemed significant by the investigator. In addition, recordable outcomes requiring positive-pressure ventilation, central venous access, intubation, chest compressions, IV vasopressors, IV vasodilators, IV anti-arrhythmics, IV fluid bolus, and/or emergency dialysis or resulting in death will be collected.

Available data obtained as part of SOC management will include physical examinations, vital signs, fluid intake and urine output, ECGs, clinical laboratory data, and results of chest x-rays. Data regarding the subject's chief complaint upon admission to the ED, the possible cause of the subject's hyperkalemia, and admitting and discharge diagnosis will be recorded; the subject's overall discharge summary will also be collected. As applicable, dates and times will be recorded for the following: ED admission, hospital admission, intensive care unit admission, observation unit admission, step down admission, regular floor admission, discharge (from any and all admissions), dialysis, Do Not Resuscitate order, death, and any other event deemed significant by the investigator. If feasible, billing information and/or Diagnosis-Related Group (DRG) codes and/or Ambulatory Payment Classifications (APC) associated with the ED visit and interventions/treatments will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* 18 years of age or older.
* Hyperkalemia confirmed in the ED (documented SOC potassium value ≥ 5.5 mmol/L; after 50 subjects with a SOC potassium value < 6.0 mmol/L have been enrolled, this criterion increases to ≥ 6.0 mmol/L).

Exclusion Criteria:

* Subjects who, in the opinion of investigator, are unable to perform the tasks associated with the protocol.
* Subjects participating in another clinical study (eg, investigational agent), which could impact this study.
* Subjects who previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with moderate to severe hyperkalemia [a Standard of Care (SOC) potassium value ≥ 5.5 mmol/L] admitted to the ED will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Absolute change in potassium over 4 hours following the initial intervention/treatment for hyperkalemia. | 4 hours
  If no intervention/treatment for hyperkalemia during ED admission, then change over 4 hours following baseline potassium measurement.

SECONDARY OUTCOMES:
Choice of intervention/treatment | 4 hours
  Changes in study-related potassium following intervention/treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Chair — ZS Pharma, Inc.
Locations (8):
- United States (8):
  - Montgomery, Alabama
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Stony Brook, New York
  - Columbus, Ohio
  - Temple, Texas

REFERENCES:
- See also: Clinical Summary — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14631&filename=ZS%20007%20Clinical%20Summary.pdf